CLINICAL TRIAL: NCT05552053
Title: Resources, Inspiration, Support and Empowerment (R.I.S.E.) for Black Pregnant Women
Brief Title: Resources, Inspiration, Support and Empowerment (RISE) for Black Pregnant Women
Acronym: RISE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of California, Los Angeles (Other); Maternal Mental Health NOW (Unknown); Candlelit Therapy (Unknown)
Responsible Party: Principal Investigator, Eynav Accortt, Clinical Psychologist, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00002283; 1R21MD017396-01A1 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related; Pregnancy Complications; Pregnancy, High Risk; Depression; Depression, Postpartum; Perinatal Depression; Anxiety; Anxiety in Pregnancy; Stress, Psychological; Racism; Discrimination, Racial; Inflammation
MeSH Terms: conditions — Pregnancy Complications; Depression; Depression, Postpartum; Anxiety Disorders; Stress, Psychological; Racism; Inflammation

STUDY DESIGN:
Intervention Model Description: This RCT will examine the clinical effectiveness of the Candlelit Care mobile health intervention at reducing mental and physical health risk compared to the standard Maternal Wellness Self-Help (MWSH) mobile health application.
  Hypothesis 1a: Compared to a standard of care control group (N=75), Black pregnant women (N=75) randomized to MWSH + Candlelit Care and structured postpartum follow up will have reduced rates of APOs and PMADs.
  Hypothesis 1b: Among women diagnosed with PMADs, participants in the intervention group will have an increase in adherence to recommended postpartum mental health treatment. They will also report increased self-advocacy skills, increased communication with providers, and reduced levels of perceived medical discrimination.
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the investigators will know which group women have been randomized to. The care provider must know, in order to properly assist with use of the mobile health application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Wellness Self Help (MWSH) Application (Active Comparator): The Maternal Wellness Self Help (MWSH) app was created to help individuals to identify and manage perinatal depression and anxiety. The app is designed is to meet the emotional needs of those who are pregnant, want to become pregnant or have given birth. This psycho-educational app informs and normalizes the range of emotional responses throughout the reproductive journey. By learning about perinatal mental health, this app hopes to empower patients to understand and name their experiences.
  Interventions: Device: MWSH
- MWSH plus Candlelit Care (Experimental): Candlelit Care is a virtual perinatal mental health application that builds on cognitive behavioral therapy (CBT) to provide Black, Indigenous and POC women and birthing parents access to culturally affirming mental health support during pregnancy. Driven by an integrated care team, women have access to self-guided therapeutic tools, peer coaching and education about perinatal mood disorders as a primary resource. This convenient and trauma informed app allows parents to see if their mental health symptoms warrant further treatment in a secure setting. The app also provides education of role transitions, discussion of types of interpersonal conflicts common around childbirth (including racial discrimination) and techniques for resolving them, and role-playing with feedback from other parents during groups. The goals are to improve self-advocacy skills; patient communication with medical providers and provide a support network with other Black pregnant women.
  Interventions: Device: MWSH plus Candlelit Care

INTERVENTIONS:
Device: MWSH plus Candlelit Care — Candlelit Care is a virtual perinatal mental health application that builds on cognitive behavioral therapy (CBT) to provide Black, Indigenous and POC women and birthing parents access to culturally affirming mental health support during pregnancy. Driven by an integrated care team, women have access to self-guided therapeutic tools, peer coaching and education about perinatal mood disorders as a primary resource. This convenient and trauma informed app allows parents to see if their mental health symptoms warrant further treatment in a secure setting. The app also provides education of role transitions, discussion of types of interpersonal conflicts common around childbirth (including racial discrimination) and techniques for resolving them, and role-playing with feedback from other parents during groups. The goals are to improve self-advocacy skills; patient communication with medical providers and provide a support network with other Black pregnant women.
  Arms: MWSH plus Candlelit Care
Device: MWSH — The Maternal Wellness Self Help (MWSH) app was created to help individuals to manage perinatal depression and anxiety. The app is designed is to meet the emotional needs of those who are pregnant, want to become pregnant or have given birth. This psycho-educational app informs and normalizes the range of emotional responses throughout the reproductive journey. By learning about perinatal mental health, this app hopes to empower patients to understand and name their experiences.
  Arms: Maternal Wellness Self Help (MWSH) Application

SUMMARY:
Perinatal Mood and Anxiety Disorders (PMADs) encompass a range of mental health disorders that occur during pregnancy and up to one year postpartum. Approximately 13% of women experience PMADs. This rate doubles for those with adverse perinatal outcomes (APO) and triples in Black women. Recent research points to racism as one significant source of these health disparities. Cultural adaptations to improve communication with providers decrease rates of depression in minority patients as well as improve adherence to treatment, insight and alliance. Discrimination stress and worries about experiencing medical consequences are thought to increase systemic inflammation, a mechanism known to drive mental and physical symptoms. Inflammation has been implicated in both PMADs and APO, suggesting a shared underlying etiology. Evidence from our work suggests that inflammation contributes to the pathophysiology of PMADs. The proposed pilot randomized control trial will allow the investigators to build on promising preliminary results and identify whether our culturally relevant mobile Health (mHealth) intervention is effective in improving outcomes among Black pregnant women randomized to the intervention compared to a control group. The culturally relevant modules include building communication and self-advocacy skills and provide a support network. The primary objective of this research is to provide guidance for clinical care of Black women during the perinatal period, with the goal to improve mental health and physical health outcomes. A secondary goal is to examine novel inflammatory signatures that change as a function of the intervention to reduce PMADs in this population. As inflammation may be diagnostic of PMADs, identification of its role may shed light of potential intervention targets and provide critical knowledge to improve women's long-term health. PMAD symptoms will be assessed prospectively in 150 Black pregnant women, half of whom will be randomized to receive the culturally relevant mHealth intervention. The investigators hypothesize that women in the intervention group will have reduced rates of PMADs and APOs, an increase in adherence to mental health treatment and will report increased self-advocacy skills, increased communication with providers, and reduced levels of discrimination related stress. Participants will also have improved biological risk indicators including lower circulating C-reactive protein and a transcription profile of differentially expressed inflammatory genes, marked by a decreased activity of inflammatory transcription factors from blood spots. Given the high burden of both PMADs and APOs among Black mothers and the numerous consequences on maternal and child outcomes, it is imperative that investigators develop and implement effective interventions, and test the biological mechanisms that might drive these effects. This work is interdisciplinary, building on a network of community advocates to implement a novel mHealth intervention informed by real world experiences designed to enhance self-advocacy, reduce stress and prevent adverse outcomes

DETAILED DESCRIPTION:
Perinatal mood and anxiety disorders (PMADs) are a leading complication of childbirth with a national prevalence rate of 13%.1-3 This rate triples among Black mothers in Los Angeles (36%)4 who are less likely to receive mental health treatment, particularly during COVID-19.5 Negative impacts of untreated depression or anxiety during pregnancy, coupled with and/or compounded by racism, can include gestational diabetes, prematurity, small gestational age and low birth weight6 - adverse perinatal outcomes (APO) that already disproportionately burden Black women.7-12 The stress of discrimination, worries about adverse outcomes, and APO consequences are thought to increase systemic inflammation,13,14 a mechanism driving mental and physical symptoms. Additionally, research shows that Black patients experience worse communication with their physicians than their white counterparts.15-17 Cultural adaptations to improve communication with providers decrease rates of depression in minority patients18 and improve adherence to insight and alliance.19 In addition to communication barriers and despite recent national recommendations and state laws,20-22 fewer than one in four Los Angeles women receive PMAD screening or education during their prenatal, postpartum or well-child medical visits.23 Based on our team's preliminary data, even when screened many women of color do not respond openly to these questions and few are connected to relevant care.24,25 Finally, a consistent problem is the lack of postpartum follow up for medical and mental health concerns.26 Together the result is a gross lack of referral to appropriate postpartum mental health care and mobile health (mHealth) apps could bridge this divide.

Our community partner Maternal Mental Health NOW developed a Maternal Wellness Self-Help (MWSH) Application that provides PMAD psychoeducation, stress management techniques and tailors a self-help plan for its 700+ users. Given the racial disparities in maternal health it became apparent that content directly addressing the unique cultural needs of Black women was critically needed. Therefore the investigators partnered with Candlelit Therapy, a culturally-relevant, virtual-first telemedicine provider focused on health equity and providing culturally competent behavioral healthcare to change the way Black mothers access perinatal mental healthcare online and get primary care. Candlelit Therapy has developed our intervention, Candlelit Care, which includes three new culturally relevant modules for Black pregnant women to improve (1) self-advocacy skills (2) patient communication with medical providers and (3) provide a support network with other Black pregnant women. In this proposed pilot randomized control trial (RCT) women will be randomized to either the active standard of care control (MWSH) or the standard of care plus the additional modules (MWSH + Candlelit Care).

The proposed pilot RCT will allow the investigators to build on the established MWSH app by adding Candlelit Care, which are culturally relevant modules and to test if it is effective in improving perinatal mental and physical health outcomes among Black Women randomized to the intervention compared to the standard of care control group. Women randomized to the intervention will also have postpartum follow up at regular intervals including additional PMAD screening by a licensed clinician who will provide patient navigation to mental health and/or medical care, if needed. The overarching objective of this research is to improve clinical care of Black women during the perinatal period, with the goal to improve mental health and physical health outcomes. A secondary goal is to identify a plausible biological mechanism through which this intervention is operating.

AIM 1: This RCT will examine the clinical effectiveness of the MWSH App + Candlelit Care intervention at reducing mental and physical health risk. Hypothesis 1a: Compared to a standard of care control group who only receive the MWSH App (N=75) Black pregnant women (N=75) who are randomized to the intervention (MWSH + Candlelit Care), and structured postpartum follow up will have reduced rates of APOs and PMADs. Hypothesis 1b: Among women diagnosed with PMADs, participants in the intervention group will report increased self-advocacy skills, increased communication with providers, and reduced levels of discrimination stress. Participants will also have an increase in adherence to recommended postpartum mental health treatment.

AIM 2: Investigate the physiological mechanisms involved. Hypothesis 2: Black pregnant women who are randomized to MWSH + Candlelit Care (n=25) will have lower circulating inflammation (hs-CRP), and a transcription profile of differentially expressed inflammatory genes, marked by a decreased activity of inflammatory transcription factors NFкB, CREB and JUN compared to the standard MWSH (n=25),

Given the burden of both APOs and PMADs among Black mothers and the numerous consequences on maternal and child outcomes, it is imperative that investigators develop and implement targeted and effective PMAD interventions, and test the biological mechanisms that might drive these effects. This work is translational, builds on a network of community advocates and established clinical providers to implement a novel mHealth intervention informed by real world experiences designed to enhance self-advocacy, reduce stress, and prevent adverse outcomes. This pilot RCT will inform a larger multi-site clinical trial to address mental health disparities in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Pregnant Black individuals, at least 18 years of age
4. English speaking
5. Access to a tablet, smartphone, or computer capable of running the apps

Exclusion Criteria:

1. Psychosis
2. Perinatal loss
3. Individuals outside of the US

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | 6 months - 1 year
  Reduced symptoms of depression assessed by the Edinburgh Postnatal Depression Scale (EPDS)
Anxiety symptoms | 6 months - 1 year
  Reduced symptoms of anxiety assessed by the Overall Anxiety Severity and Impairment Scale (OASIS)
PTSD Symptoms | 6 months - 1 year
  Reduced symptoms of post-traumatic stress symptoms assessed by the Impact of EVents Scale (IES)

SECONDARY OUTCOMES:
Communication | 6 months - 1 year
  Increased communication with providers assessed by the Communication Assessment Tool (CAT)
Self-Advocacy | 6 months - 1 year
  Improved self-advocacy skills assessed by the Patient Self-Advocacy Scale (PSAS)
Discrimination stress | 6 months - 1 year
  Reduced levels of discrimination stress assessed by the Discrimination in Medical Settings (DMS) Scale.

OTHER OUTCOMES:
Inflammation | 6 months - 1 year
  Lower circulating inflammation (hs-CRP), and a transcription profile of differentially expressed inflammatory genes, marked by a decreased activity of inflammatory transcription factors NFкB, CREB and JUN.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai, Los Angeles, California, United States